CLINICAL TRIAL: NCT05557565
Title: A Single-arm, Open, Multicenter Phase II Trial to Evaluate the Efficacy and Safety of QL1706 in Patients With Recurrent or Metastatic Cervical Cancer
Brief Title: A Phase II Trial to Evaluate the Efficacy and Safety of QL1706 in Patients With Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-206
Record Dates: First submitted 2022-09-20; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 injection (Experimental): The dosage of QL1706 is 5.0 mg/kg, and QL1706 is administered every 3 weeks (Q3W) by intravenous infusion
  Interventions: Drug: QL1706

INTERVENTIONS:
Drug: QL1706 — The dosage of QL1706 is 5.0 mg/kg, and QL1706 is administered every 3 weeks (Q3W) by intravenous infusion

SUMMARY:
This is a single-arm, open-label, multicenter, phase II trial to evaluate the efficacy and safety of QL1706 in patients with recurrent or metastatic cervical cancer.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter, phase II trial to evaluate the efficacy and safety of QL1706 in patients with recurrent or metastatic cervical cancer who have failed at least first-line platinum-containing standard therapy.

The study was divided into screening period/baseline, treatment period, and post-treatment follow-up period. Efficacy evaluation and safety monitoring should be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject will participate voluntarily and sign the informed consent form.
* Female, aged ≥18 years when signing the informed consent form.
* Recurrent or metastatic cervical cancer (pathological types include squamous cell carcinoma, adenocarcinoma) which is not suitable for radical treatment such as surgery and radiotherapy.
* At least one measurable lesion is needed.
* The Eastern Collaborative Oncology Group (ECOG) physical status score was 0 or 1.
* Adequate reserves of organ function is needed.

Exclusion Criteria:

* Active autoimmune disease.
* Central nervous system (CNS) metastasis.
* Concomitant diseases such as cardiovascular and cerebrovascular diseases.
* Fistula of female genital tract.
* Diseases for which systemic corticosteroids or other immunosuppressive agents are planned to be used during the study treatment.
* Previous recipients of immune checkpoint inhibitors.
* Received systemic antitumor drugs such as chemotherapy and targeted therapy within 4 weeks before the first use of the experimental drug; Received proprietary Chinese medicine with anti-tumor indications within 2 weeks before the first use of the experimental drug.
* Received radical concurrent chemoradiotherapy or adjuvant chemoradiotherapy within 12 weeks before the first use of the investigational drug; Received palliative radiotherapy (e.g., reductive radiotherapy for pain or bleeding) or other local treatments (e.g., radiofrequency ablation, transarterial chemoembolization, etc.) within 2 weeks before the first use of the investigational drug.
* History of immunodeficiency.
* History of allogeneic hematopoietic stem cell transplantation or organ transplantation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The Overall Response Rate (ORR) assessed by the Independent Image Review Board (IRC) | Every 6 weeks, from the date of enrollment until the date of the last time that tumor imaging and assessment of disease has been done, assessed up to 2 years
  The ORR assessed by the Independent Image Review Board (IRC) according to RECIST V1.1

SECONDARY OUTCOMES:
The Overall Response Rate (ORR) assessed by the investigator according to RECIST V1.1 | Every 6 weeks, from the date of enrollment until the date of the last time that tumor imaging and assessment of disease has been done, assessed up to 2 years
  The ORR assessed by the investigator according to RECIST V1.1
The Disease Control Rate (DOR) assessed by the Independent Image Review Board (IRC) and the investigator | Every 6 weeks, from the date of enrollment until the date of the last time that tumor imaging and assessment of disease has been done, assessed up to 2 years
  The DOR assessed by the Independent Image Review Board (IRC) and the investigator according to RECIST V1.1
The Progression-free survival (PFS) assessed by the Independent Image Review Board (IRC) and the investigator | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the last QL1706 injection has been administered.
  The PFS assessed by the Independent Image Review Board (IRC) and the investigator according to RECIST V1.1
Overall survival | From date of enrollment until the date of death from any cause or date of lost to visit, assessed up to 2 years after the last QL1706 injection has been administered.
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No